CLINICAL TRIAL: NCT04614220
Title: The Correlation Between Family Member Presence and The Consent for Regional Anaesthesia for Cesarean Section of Primigravida: A Prospective Observational Study
Brief Title: The Correlation Between Family Member Presence and The Consent for Regional Anaesthesia for Caesarean Section
Acronym: BSU
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mahmoud Hussein Bahr, Lecturer in Department of Anaesthesia , surgical ICU and pain management (Faculty of medicine), Beni-Suef University
Other Study IDs: FMBSUREC/04102020/ Bahr
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Acceptability of Health Care
Keywords: Caesarean Section; Regional anaesthesia; Consent
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Presence of Family member — The correlation between presence of the Family member and the consent for regional anaesthesia for Caesarean Section

SUMMARY:
Patient's safety and satisfaction are major concerns of anesthesiologists and obstetricians. According to evidence guidelines, and quality markers, regional anesthesia is preferred over general in obstetric surgery. Already a high level of anxiety is present in obstetric patients preoperatively.

DETAILED DESCRIPTION:
Hospital anxiety is commonly encountered, and it is reported to be seen in 60%-80% of patients who undergo surgery. There are many causes of preoperative anxiety including fear of death due to anesthesia or surgical procedure and fear of preoperative or postoperative pain.

Preoperative anxiety varies according to the patient's age, gender, educational status, history of previous operations, and medical status as well as the type of surgery and type of anesthesia. Patient's safety and satisfaction are major concerns of anesthesiologists and obstetricians. According to evidence guidelines, and quality markers, regional anesthesia is preferred over general in obstetric surgery. Already a high level of anxiety is present in obstetric patients preoperatively.

The anxious patients tend to prefer general anesthesia (GA) for cesarean section (CS). The patient refusal is the main contraindication for applying spinal anesthesia (SA) during CS. The anxiety can be reduced variably by non-pharmacologic and pharmacologic methods including preoperative visit, information, and music, listening to Holy Quran recitation, hypnosis, nitrous oxide, and benzodiazepines. Intravenous sedation can control the anxiety in 90% of patients subjected to spinal procedures. While the evidence supports the benefits of procedural sedation for distressed, anxious pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* primi gravida Patients aging 20_40 years, ASA physical status I undergoing elective CS •

Exclusion criteria:

High risk pregnancy eg: pre eclampsia Absolute contra indiction for SA eg: severe anaemia Emergent CS. Patients with previous exposure to anaesthesia ( spinal or general ). Patients with educational level more than high school.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Caesarean Section
Study Population: 110 primi gravida Patients aging 20_40 years, ASA physical status I undergoing elective CS •
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Acceptance rate to spinal anaethesia during CS | Preoperative .
  Questionnaire : The first decision for anesthesia, either spinal or general, will be recorded.
  Then, patients who refuse SA and prefer general anesthesia (GA) will be consulted again as regards SA with presence of close relative for comfortable spinal procedure. Their last choice is the second decision that determines the final type of anesthesia to be implemented.
Anxiety score by the visual analogue score (VAS). | Preoperative
  the visual analog score (VAS) from 0- 10, where 10 is the maximum anxiety level
Satisfaction rating scale | 6 hours Postoperative
  Scale ( 1 - 10 )
  1is the lowest satisfaction 10 is the best satisfaction

SECONDARY OUTCOMES:
AGE | Preoperative
  age per years
heart rate (beat/min) | Preoperative
  heart rate (beat/min)
Mean arterial blood pressure MAP (mmHg) | Preoperative
  Mean arterial blood pressure MAP (mmHg)
peripheral oxygen saturation (Spo2) | Preoperative
  peripheral oxygen saturation (Spo2)
WEIGHT | Preoperative
  weight per kilograms
Height | Preoperative
  Height per centimeter

CONTACTS AND LOCATIONS:
Overall Officials: Amira F Elgamel, Lecturer, Study Director — Faculty of medicine.Beni-suef university
Locations (1):
- Faculty of medicine.Beni-suef university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The surgeon and the anesthetist will discuss the exclusion criteria, and then discuss the information about spinal and general anesthesia with the illegible patients. The first decision for anesthesia, either spinal or general, will be recorded.
  Then, patients who refuse SA and prefer general anesthesia (GA) will be consulted again as regards SA with presence of close relative for comfortable spinal procedure. Their last choice is the second decision that determines the final type of anesthesia to be implemented. The acceptance rate of SA with presence of close relative will be the primary outcome. A written consent will be taken. The number of crying patients and anxiety causes will be documented just before SA. The anxiety score will be assessed by the visual analog score (VAS) from 0- 10, where 10 is the maximum anxiety level .
Supporting Information: Study Protocol, ICF
Time Frame: 3 months
Access Criteria: drmahmoudbahr@gmail.com
URL: https://www.bsu.edu.eg/home.aspx?lang=en